CLINICAL TRIAL: NCT01579734
Title: The HOT Study: Hormone Replacement Therapy Opposed by Low Dose Tamoxifen. A Phase III Trial of Breast Cancer Prevention With Low Dose Tamoxifen in HRT Users.
Brief Title: Phase III, Randomized, Double Blind Trial Low Dose Tamoxifen Versus Placebo in Hormone Replacement Therapy (HRT) Users
Acronym: HOT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IEO S51/200
Record Dates: First submitted 2012-01-24; First posted 2012-04-18 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: breast cancer chemoprevention postmenopause
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1 tablet day for 5 years
  Interventions: Drug: Placebo
- Tamoxifen (Active Comparator): Tamoxifen 5 mg, (1 tablet) day for 5 years
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — 1 tablet, 5 mg / day for 5 years
  Other Names: Nolvadex, Istubal, Valodex
  Arms: Tamoxifen
Drug: Placebo — 1 tablet day for 5 years
  Arms: Placebo

SUMMARY:
The propose of this trial is to assess the effect of low dose tamoxifen for breast cancer prevention in HRT (Hormone Replacement Therapy)users.

DETAILED DESCRIPTION:
While life expectancy has grown by approximately 30 years in the last century in western countries, the age at menopause has increased by 2-3 years only. Thus, women are exposed to postmenopausal symptoms and disorders related to estrogens drop for a considerable period of their lifetime. The management of these frequent disorders is an important public health issue. Although recent data from the WHI randomized trial have demonstrated that late postmenopausal women (mean age 63.3 years) taking oral conjugated equine estrogens and medroxyprogesterone acetate in a continuous combined regimen for prevention of coronary heart disease have an increased risk of developing cardiovascular disease and breast cancer, there is no question that treatment of menopausal symptoms with HRT (Hormone Replacement Therapy) in younger women aged around 50 years is a clinically beneficial treatment. This is even truer for women who enter menopause earlier than 45 years. It is prudent not to extend the results of the WHI trial, as such, to other forms of HRT preparations, routes, dosages and regimens or to early postmenopausal women with no apparent risk factors for CVD. Recently data from a non-randomized study, the Million Women Study, have suggested that oral combined regimens are associated with an increased and that transdermal estradiol does not increase more than oral treatment, and in general may be less harmful: for instance, transdermal estradiol has no effect on vascular inflammatory markers in contrast to the increase observed with oral CEE (conjugated equine estrogens). Notably, more recent data on the estrogens-alone group of the WHI trial show a lower breast cancer risk than the combination, suggesting a important role of progestin in the risk, and a significant reduction in colon cancer.

The increased risk of developing breast cancer, mostly estrogens receptor positive, particularly with the combination of estrogens and progestin, has been associated with an increased expression of estrogens receptors in the healthy breast tissue, thus leading to an enhanced sensitivity to the estrogens signal. Moreover, reproductive factors such as early menarche and delayed pregnancy are also associated with a higher risk of estrogens receptor (ER) positive breast cancer. Thus, the addition of a SERM may reduce the hormone growth-promoting effect on the breast gland. Tamoxifen has been investigated in four large cooperative phase III trials for breast cancer prevention in at-risk women. While the preliminary results of the Italian Tamoxifen Prevention Study in hysterectomized women showed no difference between arms, a recent update after 7 years of follow-up suggests that the combination of HRT and tamoxifen has a favorable effect and might even be synergistic. At a mean observation time of 81 months, a 25% reduction of breast cancer was noted in the tamoxifen arm compared with placebo (45 versus 34 events, Hazard Ratio, HR= 0.75, 95% CI, 0.48-1.18). While there is no difference in the subset of women who never took HRT before or during the trial (HR=1.01, 95% CI, 0.60-1.70), women, who at some point before or during the study, had ever taken HRT (n=1584) had fewer breast cancers in the tamoxifen arm (6 on tamoxifen versus 17 on placebo, HR=0.35, 95% CI, 0.14-0.89). Among the women continuously on HRT during the trial (n= 754), breast cancer events were 3 for women on tamoxifen versus 11 for those on placebo, respectively (HR=0.30, 95% CI, 0.08-1.06). Notably, 76.9% of HRT users received transdermal unopposed ERT and further 6.5% took transdermal ERT combined with progestins. Importantly, recent result from the IBIS I trial indicate that there is no evidence that HRT use affects the tamoxifen benefit. Recent studies suggest that the standard dose of tamoxifen may be reduced to one quarter (5 mg day) without significant loss of its beneficial effects on circulating biomarkers, mostly reflecting cardiovascular risk. Moreover, the efficacy of doses as low as one twentieth of the standard 20 mg/day dose on breast cancer cell proliferation has been recently shown. Since the endometrial effect of tamoxifen is dependent on treatment duration and dose, a dose reduction might reduce the risk of endometrial malignancies, while retaining its preventive efficacy. On the other hand, the addition of HRT containing progestins could further minimize the risk of endometrial cancer associated with tamoxifen. Moreover, estrogen should reduce the incidence of vasomotor and uro-genital symptoms, which are a major reason for tamoxifen withdrawal in prevention studies. In the NSABP trial, women aged 50 or younger demonstrated no significantly increased incidence of severe adverse events, including endometrial cancer and, even more importantly, venous thromboembolic events (VTE). One possible explanation for the lack of severe toxicity in premenopausal women is the concomitant presence of adequate circulating estrogens levels which prevent tamoxifen from acting as an estrogens agonist on these target tissues. Notably, in the IBIS I trial, no significant excess of endometrial cancer and VTE was noted in the women on HRT who were allocated to tamoxifen compared to placebo.

The above background provides the rationale for a phase III chemoprevention trial in postmenopausal healthy women HRT users and Tamoxifen: the HOT Study (Hormone replacement therapy Opposed by low dose Tamoxifen).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women candidates to HRT for control of menopausal symptoms or prevention of postmenopausal disorders. women currently undergoing HRT for any duration; (women off HRT for 1 year or longer are considered de novo users);
* negative bilateral mammography (within the last 6 months);
* written informed consent.

Exclusion Criteria:

Any type of malignancy, with the exclusion of CIN and non-melanoma skin cancer;

* active proliferative disorders of the endometrium such as atypical hyperplasia, history of active endometriosis, unresected polyps, symptomatic myomata;
* alterations of metabolic, liver, renal and cardiac grade 2 function (NCI criteria grade 2 or higher);
* any type of retinal disorders, severe cataract and glaucoma;
* presence of significant risk factors for venous events, including immobilization within the last 3 months for longer than 2 weeks following surgery or trauma, history of estrogen-associated and "sine causa" superficial phlebitis, deep venous thrombophlebitis or other significant VTE (pulmonary embolism, stroke, etc.);
* use of tamoxifen, raloxifene or other SERMs within the last 4 weeks;
* anticoagulant therapy in progress (heparin or dicoumarol);
* active infections;
* severe psychiatric disorders or inability to comply to the protocol procedures; any other factor that at the investigator's discretion contraindicates the use of either tamoxifen or HRT.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1884 (Actual)
Dates: Start 2002-03; Primary Completion 2018-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
breast cancer incidence | 10 years
  The primary objective is to assess if tamoxifen at a low dose reduces the incidence of breast cancer in healthy postmenopausal women undergoing or willing to initiate hormone replacement therapy (HRT), including the women who will eventually withdraw HRT during the 5 year intervention period and additional 5 years of follow up.

SECONDARY OUTCOMES:
Incidence of adverse events | 10 years
  Incidence of: other non-invasive breast disorders (i.e., LCIS, atypical hyperplasia) All other cancers (with special reference to endometrial cancer, colorectal cancer, ovarian cancer and melanoma).
  Bone fractures Cardiovascular events Venous thromboembolic events Clinically manifest cataract Overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Veronesi, MD, Study Chair — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy